CLINICAL TRIAL: NCT02702505
Title: Success and Color Stability of MTA Pulpotomized Primary Molars: an RCT
Acronym: MTA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas A & M University Baylor College Of Dentistry (Other)
Responsible Party: Principal Investigator, Carolyn A. Kerins DDS, Associate Professor and Graduate Program director, Texas A & M University Baylor College Of Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 072015-041
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Reversible Pulpitis; Dental Pulp Diseases
Keywords: Pulp; pulpotomies; mineral trioxide aggregate
MeSH Terms: conditions — Dental Pulp Diseases | interventions — ProRoot MTA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeoMTA (Experimental): The new formulation of MTA (does not contain bismuth oxide) will be used in one tooth receiving a pulpotomy to determine if the color of the tooth changes over time. The new formulation has received the Food and Drug Administrations 510(k) substantial equivalence clearance for Class II dental materials and is equivalent to its MTA predicate (ProRoot, Dentsply Tulsa Dental, Tulsa, OK, USA).19
  Interventions: Biological: NeoMTA
- ProRoot MTA (Other): Control group. This group will receive the old formulation of MTA in the pulpotomy and the tooth will receive a full coverage stainless steel crown restoration.
  Interventions: Other: ProRoot MTA

INTERVENTIONS:
Biological: NeoMTA — A new formulation of MTA was developed in which bismuth oxide was omitted
  Arms: NeoMTA
Other: ProRoot MTA — Control group
  Arms: ProRoot MTA

SUMMARY:
Mineral trioxide aggregate has been previously FDA approved as an endodontic filler. Its use in vital teeth has demonstrated significant color change post-treatment leaving it ineffective for esthetic use..

The new formulation will be tested to see if has the same effect.

DETAILED DESCRIPTION:
This randomized control, split-mouth trial will use 50 pediatric subjects selected from the patient population in the pediatric dental clinics at Baylor College of Dentistry and in select faculty private practices. The study will use a within-subject control design whereby one tooth will be treated with a pulpotomy using the new formulation of MTA (NeoMTA Plus, Avalon Biomed Inc., Bradenton, FL, USA) and restored with a multi-surface composite, and the other tooth with an MTA pulpotomy and restored with a SSC; thus, approximately 50 teeth will be treated for each treatment group. The restoration type will be randomized as to which side will receive the SSC or composite using sealed, opaque envelopes. Approximately 50 subjects will be needed for the study in order to elicit any significant findings as demonstrated by a power analysis from a similar study.

ELIGIBILITY:
Inclusion Criteria:

* • Children between the ages of 2 ½ and 8 years of age

  * Patient must have two, contralateral primary molars that are matched for type of molar (first or second), size of carious lesion (same level of approximation of carious lesion to the pulp), and arch (maxillary or mandibular) that are treatment planned for a pulpotomy
  * The teeth selected for the study must be vital and asymptomatic both clinically and radiographically or only display symptoms consistent with reversible pulptitis
  * The teeth selected for the study must be anticipated to be retained in the mouth for at least two years
  * Each patient must have an updated medical history form in the dental record, be examined by the operator, and be classified as ASA I or II (in good general health)

Exclusion Criteria:

* Teeth with a history of spontaneous pain
* Teeth with radiographic evidence of internal or external resorption, intraradicular or periapical bone loss, loss of lamina dura, or widening of the periodontal ligament space

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Color stability | 2 years
  Dental intraoral photographs will evaluated
Internal resorption | 2 years
  Dental radiographs will be evaluatedresorption
external resorption | 2 years
  Dental radiographs will be evaluated resorption
Bone loss | 2 years
  Dental radiographs will be evaluated for intraradicular or periapical bone loss
Widening of periodontal ligament space | 2 years
  Dental radiographs will be evaluated for widening of the PDL space

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A Kerins, DDS, PhD, Principal Investigator — Texas A & M University Baylor College Of Dentistry
Locations (1):
- Texas A & M University Baylor College of Dentistry, Dallas, Texas, United States

REFERENCES:
- [Background] Agamy HA, Bakry NS, Mounir MM, Avery DR. Comparison of mineral trioxide aggregate and formocresol as pulp-capping agents in pulpotomized primary teeth. Pediatr Dent. 2004 Jul-Aug;26(4):302-9. PMID 15344622
- [Background] Farsi N, Alamoudi N, Balto K, Mushayt A. Success of mineral trioxide aggregate in pulpotomized primary molars. J Clin Pediatr Dent. 2005 Summer;29(4):307-11. doi: 10.17796/jcpd.29.4.n80t77w625118k73. PMID 16161395
- [Background] Holan G, Eidelman E, Fuks AB. Long-term evaluation of pulpotomy in primary molars using mineral trioxide aggregate or formocresol. Pediatr Dent. 2005 Mar-Apr;27(2):129-36. PMID 15926290
- [Background] 4. Jabbarifar SE, Khademi D, Ghasemi D. Success rates of formocresol pulpotomy versus mineral trioxide aggregate in human primary molar tooth. J Res Med Sci 2004; 9(6)L 55-8.
- [Background] Peng L, Ye L, Tan H, Zhou X. Evaluation of the formocresol versus mineral trioxide aggregate primary molar pulpotomy: a meta-analysis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Dec;102(6):e40-4. doi: 10.1016/j.tripleo.2006.05.017. Epub 2006 Sep 26. PMID 17138165
- [Background] Farooq NS, Coll JA, Kuwabara A, Shelton P. Success rates of formocresol pulpotomy and indirect pulp therapy in the treatment of deep dentinal caries in primary teeth. Pediatr Dent. 2000 Jul-Aug;22(4):278-86. PMID 10969431
- [Background] Guelmann M, Fair J, Bimstein E. Permanent versus temporary restorations after emergency pulpotomies in primary molars. Pediatr Dent. 2005 Nov-Dec;27(6):478-81. PMID 16532888
- [Background] Holan G, Fuks AB, Ketlz N. Success rate of formocresol pulpotomy in primary molars restored with stainless steel crown vs amalga. Pediatr Dent. 2002 May-Jun;24(3):212-6. PMID 12064493
- [Background] Caceda JH. The use of resin-based composite restorations in pulpotomized primary molars. J Dent Child (Chic). 2007 May-Aug;74(2):147-50. PMID 18477438
- [Background] Cehreli ZC, Cetinguc A, Cengiz SB, Altay AN. Clinical performance of pulpotomized primary molars restored with resin-based materials. 24-month results. Am J Dent. 2006 Oct;19(5):262-6. PMID 17073200
- [Background] Guelmann M, Bookmyer KL, Villalta P, Garcia-Godoy F. Microleakage of restorative techniques for pulpotomized primary molars. J Dent Child (Chic). 2004 Sep-Dec;71(3):209-11. PMID 15871455
- [Background] Guelmann M, McIlwain MF, Primosch RE. Radiographic assessment of primary molar pulpotomies restored with resin-based materials. Pediatr Dent. 2005 Jan-Feb;27(1):24-7. PMID 15839391
- [Background] Hutcheson C, Seale NS, McWhorter A, Kerins C, Wright J. Multi-surface composite vs stainless steel crown restorations after mineral trioxide aggregate pulpotomy: a randomized controlled trial. Pediatr Dent. 2012 Nov-Dec;34(7):460-7. PMID 23265162
- [Background] Maroto M, Barberia E, Planells P, Garcia Godoy F. Dentin bridge formation after mineral trioxide aggregate (MTA) pulpotomies in primary teeth. Am J Dent. 2005 Jun;18(3):151-4. PMID 16158803
- [Background] Parirokh M, Asgary S, Eghbal MJ, Stowe S, Eslami B, Eskandarizade A, Shabahang S. A comparative study of white and grey mineral trioxide aggregate as pulp capping agents in dog's teeth. Dent Traumatol. 2005 Jun;21(3):150-4. doi: 10.1111/j.1600-9657.2005.00311.x. PMID 15876326
- [Background] Holland R, de Souza V, Murata SS, Nery MJ, Bernabe PF, Otoboni Filho JA, Dezan Junior E. Healing process of dog dental pulp after pulpotomy and pulp covering with mineral trioxide aggregate or Portland cement. Braz Dent J. 2001;12(2):109-13. PMID 11445912
- [Background] American Academy on Pediatric Dentistry Clinical Affairs Committee-Pulp Therapy subcommittee; American Academy on Pediatric Dentistry Council on Clinical Affairs. Guideline on pulp therapy for primary and young permanent teeth. Pediatr Dent. 2008-2009;30(7 Suppl):170-4. No abstract available. PMID 19216417
- [Background] Zurn D, Seale NS. Light-cured calcium hydroxide vs formocresol in human primary molar pulpotomies: a randomized controlled trial. Pediatr Dent. 2008 Jan-Feb;30(1):34-41. PMID 18402097